CLINICAL TRIAL: NCT06761885
Title: Prediction of Placenta Accreta Outcome in Pregnant Woman With Placenta Previa Using (hcg_h ) as Abiomarker
Brief Title: Prediction of Placenta Accreta Outcome in Pregnant Woman With Placenta Previa Using (hcg_h ) as Abiomarkers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mahrous Fouad Mohammed, Resident of women's health Assiut University hospital, Assiut University
Other Study IDs: placenta accreta & previa
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Placenta Accreta / Percreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 74 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To check if maternal serum (hcg _h ) in second and third trimester in pregnant woman with placenta previa can predict placenta accreta at delivery or predict adverse maternal and neonatal outcome

DETAILED DESCRIPTION:
Placenta accreta was first described in 1937 by Irving et al. as failure of separation of the placenta from the uterine wall following delivery of the human fetus leading to the often used term morbid placental adherence. The condition is characterised by invasive placentation which is associated with catastrophic haemorrhage. Varied terminology has been applied to this condition; however, recent guidelines suggested that placenta accreta spectrum (PAS), which includes accreta, increta, and percreta (defined below), be used going forward.The condition is unique to human pregnancy with no animal correlate reported in the literature.The incidence of PAS has increased substantially from 0.8 per 1000 deliveries in the 1980s to 3 per 1000 deliveries in the past decade, a phenomenon attributed to a rising global caesarean section rate . PAS is associated with significant maternal morbidity and mortality, in particular, major obstetric haemorrhage and peripartum hysterectomy . Mortality rates of up to 7% have been reported to be associated with PAS . The most recent confidential inquiry into maternal mortality in the United Kingdom (MMBRACE-UK, 2017) highlighted the continued high maternal mortality associated with the condition . The most important antenatal risk factor for PAS is the number of previous caesarean sections. In the presence of low-lying placenta (placenta previa) and three previous caesarean sections, a woman would have a 61% risk of PAS. Antenatal diagnosis is a key element to improving maternal and perinatal outcome . Although dedicated ultrasound and MRI having improved antenatal diagnosis, between one half and two thirds of cases remain undiagnosed, resulting in poorer maternal outcomes.For several years, investigators have attempted to identify maternal serum biomarkers that could be used to improve the accuracy of antenatal diagnosis of PAS. The use of ultrasound and MRI in the diagnosis of PAS has been extensively reviewed elsewhere . Several placental and fetal hormones routinely used in the screening for aneuploidy have been found to be differentially expressed in the serum of women with PAS compared with those with placenta previa . HCG is a glycoprotein composed of 244 amino acids with a molecular mass of 36.7 kDa that is produced by the syncytiotrophoblast and maintains pregnancy by stimulating progesterone synthesis by the corpus luteum. A maximum level of approximately 100,000 iu/l is reached by 8-10 weeks of gestation and declines as placental steroid synthesis commences .HCG is a heterodimeric molecule composed of an alpha subunit that is identical to luteinising hormone, follicle-stimulating hormone, and thyroid-stimulating hormone and a beta (β) subunit that is unique. Proteolytic cleavage by trophoblast macrophages destabilises the molecule, thereby producing free β-hCG that is secreted into the maternal circulation . Hyperglycosylated hcg is glycosylation variant of the hormone hcg .its different molecule to regional hcg as it produced by extravillous cytotrophoblastic cell (invasive trophoblast ) its function is invasive promoter as in implantation of pregnancy where it appears to promote cell proliferation ,invasion and implantation

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* At least previous one CS
* Gestational age at second and third trimester
* Age (18:45) years

Exclusion Criteria:

* proven fetal aneuploidy in current pregnancy

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: * pregnant woman
  * At least previous one CS
  * Gestational age at second and third trimester
  * Age (18:45) years
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prediction of degree of placenta adherence by (hcg_h) and correlation intraoperative finding | 12months
  Prediction of degree of placenta adherence by (hcg_h) and correlation intraoperative finding

REFERENCES:
- See also: 1- Irving C. And Hertig A. T., A study of placenta accreta, Surgery, Gynecology & Obstetrics. (1937) 38, no. 6, 1088-1200 — https://doi.org/10.1016/S0002-9378(39)90680-0